CLINICAL TRIAL: NCT02216955
Title: Impact of Nutrition, Dietary Pattern, Obesity, Physical Activity, Depression, Diabetes, Aspirin Use and Vitamin Supplement in Colorectal Cancer in China
Brief Title: Nutrition and Lifestyle Study Cohort of Gastric Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Cancer Biology (Network)
Collaborators: Tang-Du Hospital (Other); Tianjin Union Medical Center (Other); Chengdu Medical College (Other); Beihua University (Other); Shanghai Jiao Tong University School of Medicine (Other); Second Military Medical University (Other); China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other); Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dake Chu, Dr., State Key Laboratory of Cancer Biology
Other Study IDs: cdk-201002
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
China has the largest gastric cancer patients population all over the world. Recent reports concluded nutrition status and lifestyle factors were associated with gastric cancer risk, however, the influence of nutrition and lifestyle factors on cancer outcome in gastric cancer survivors is largely unknown.The investigators will explore the impact of nutrition status, life style, dietary pattern, obesity, physical activity, depression, diabetes, aspirin use and vitamin supplement on gastric cancer outcome. The investigators will recruit approximately 50,000 patients as a prospective study cohort. During follow up, the investigators will explore the association of these factors with disease-specific survival, disease-free survival and overall survival of patients. The investigators believe that this project will facilitate the establishment of domestic nutrition and lifestyle data of gastric cancer of China, and the improvement of the quality of clinical management of patients with gastric cancer.

DETAILED DESCRIPTION:
Background - Gastric cancer incidence is increasing at an alarming rate in China. Recent studies reported that nutrition status and lifestyle factors such as dietary pattern, obesity, physical activity, depression, diabetes, aspirin use and vitamin supplement were associated cancer risk. Yet, the influence of nutrition and lifestyle factors on gastric cancer outcome (i.e. recurrence and survival) in gastric cancer survivors is largely unknown. And there is currently no large cohort studies investigated the impact of these factors on gastric cancer outcomes in China.

Objectives - Our study aims to evaluate the impact of nutrition status and lifestyle factors such as dietary pattern, tea consumption, obesity, physical activity, depression, diabetes, aspirin use and vitamin supplement on gastric cancer outcome (disease-specific survival, disease-free survival and overall survival).

Settings and methods - The study will recruit approximately 50,000 participants with gastric cancer from 12 public hospitals in China after informed consent. Appropriate questionnaires will be utilized to evaluate nutrition status and lifestyle factors such as dietary pattern, tea consumption, obesity, physical activity, depression, diabetes, aspirin use and vitamin supplement. The association of disease-specific survival, disease-free survival and overall survival with these factors will be evaluated.

Impact - To the best of our knowledge, this is the first large cohort, systematically investigation of the impact of nutrition status and lifestyle factors on gastric cancer outcome. When complete, our investigation would supply a systematical and precise understanding of the impact nutrition status and lifestyle factors on cancer out come in China.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically proven adenocarcinoma of gastric cancer.
* Patients must have a performance status of 0,1, or 2 by the Southwest Oncology Group criteria.
* Patients must have recovered from any effects of surgery.
* Evaluable disease must be present outside radiation field. At least 3 weeks must have elapsed after discontinuation of radiation therapy.
* Patients must provide a signed consent to participate in the study.
* Patients must complete all questionnaires.

Exclusion Criteria:

* Patients with a proven history of peptic ulcer disease or gastroesophageal reflux.
* History of other malignancy, except for cancers that have been treated with a curative intent and patient is without evidence of active disease.
* Unresolved bacterial infection requiring treatment with antibiotics.
* Pregnant or lactating women may not participate in the study.
* Patients known to have HIV-1 virus infection because of the undetermined effect of this chemotherapy regimen in patients with HIV-1 and the potential for serious interaction with anti-HIV medications..
* Other serious concurrent infection
* Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit about 50,000 patients with gastric cancer in 12 hospitals of China
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2009-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease-specific survival | 7 years
  Disease-specific survival is defined as the time elapsed from surgery to death due to gastric cancer. Concretely, the cause of death obtained in the follow up was classified according to ICD-10 conventions. Disease-specific deaths included those with an underlying cause attributed to ICD-10 codes C18.0-C20.0 or C26.0.

SECONDARY OUTCOMES:
Overall survival | 7 years
  Overall survival is defined as the time elapsed from surgery to the date of death from any cause

OTHER OUTCOMES:
Disease-free survival | 7 years
  Disease-free survival is defined as the time elapsed from surgery to the first occurrence of any of the following events: recurrence of gastric cancer; gastric cancer distant metastasis; development of second non-colorectal malignancy excluding basal cell carcinomas of the skin and carcinoma in situ of the cervix; or death from any cause without documentation of a cancer-related event.

CONTACTS AND LOCATIONS:
Locations (1):
- State Key laboratory of Cancer Biology, Xi'an, Shaanxi, China